CLINICAL TRIAL: NCT05747079
Title: Comparison of Immediate Versus Optional Delayed Surgical Repair for Treatment of Acute Anterior Cruciate Ligament Injury Through a Parallel, Multicentric, Pragmatic Randomized Controlled Trial
Brief Title: Immediate Versus Optional Delayed Surgical Repair for Treatment of Acute ACL Injuries
Acronym: IODA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Belgian Health Care Knowledge Centre (Unknown); Jessa Ziekenhuis Hasselt (Unknown); Centre Hospitalier Universitaire de Liege (Other); Clinique Saint-Luc Bouge (Unknown); University Hospital Brussel (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S67021
Record Dates: First submitted 2023-02-10; First posted 2023-02-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: ACL Injury
Keywords: ACL; RCT; Conservative treatment; ACL reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative treatment (Experimental): Rehabilitation and optional delayed ACL reconstruction
  Interventions: Other: Rehabilitation; Procedure: Optional delayed anterior cruciate ligament reconstruction
- Immediate ACL reconstruction (Experimental): Immediate ACL reconstruction + rehabilitation
  Interventions: Other: Rehabilitation; Procedure: Immediate anterior cruciate ligament reconstruction

INTERVENTIONS:
Other: Rehabilitation — All patients complete rehabilitation under supervision of their own physiotherapist. The investigators will provide some guidelines and criteria, but it is the physiotherapist's choice how to implement these guidelines in clinical practice.
Procedure: Optional delayed anterior cruciate ligament reconstruction — If a patient complains about persistent symptomatic instability of the knee or the inability to progress in rehabilitation, delayed surgery can be considered. ACL insufficiency induced instability in combination with a positive pivot shift and an additional MRI are needed to confirm the cause of instability.
  This surgery will not be performed within the first 12 weeks after the ACL injury.
  Arms: Conservative treatment
Procedure: Immediate anterior cruciate ligament reconstruction — No guidelines on type of ACL reconstruction will be imposed to keep the trial pragmatic. The decision of graft type and surgery technique is a clinical decision made by the orthopaedic surgeons of the participating centra.
  This surgery will be performed within 12 weeks after the ACL injury.
  Arms: Immediate ACL reconstruction

SUMMARY:
Currently, most patients with an anterior cruciate ligament injury undergo surgery. There is a general belief that surgical reconstruction is necessary to safely return to sports and to prevent early knee osteoarthritis or additional meniscus injuries. But there is insufficient scientific evidence to support this belief. Moreover, several studies show that surgical reconstruction of the cruciate ligament does not guarantee successful return to sports or the prevention of osteoarthritis and secondary meniscus injuries. Therefore, immediate surgery after an anterior cruciate ligament injury is questioned. So far, only two RCTs (KANON study and COMPARE study) have assessed this, and they could not show that immediate reconstruction is an added value (in terms of symptoms, knee function, activity level, osteoarthritis or additional meniscal injuries) compared to a conservative approach consisting of rehabilitation and late surgery for persistent knee instability.

Therefore, this additional multicenter RCT, aims to 1) verify these results and 2) to identify predictors that predict which patients in the conservative group will not require late surgery. This has not been investigated to date. It is suspected that factors such as symptoms, strength, findings on the MRI scan and psychological factors may play a role in whether or not a patient will be able to successfully rehabilitate without surgical repair.

This information is invaluable to physicians because it allows them to decide which treatment is best for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Rotational trauma to a knee that had no previous serious injury and for which medical advice was sought within 4 weeks after the injury.
* Medical diagnosis of ACL insufficiency including MRI (both partial and complete ruptures)
* Minimum of 16 years

Exclusion Criteria:

* Participant has a history of a previous ACL injury or knee surgery to the index knee
* Indication for acute surgery because of related injuries to the knee
* Female who is pregnant or plans to become pregnant in the first 4 months of the trial. Since MRI assessment cannot be performed.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2028-03-02 (Estimated)

PRIMARY OUTCOMES:
Clinical effectiveness (long-term) | 12 months post-injury
  Knee Injury and Osteoarthritis Outcome Score - Subscale Quality of Life (score between 0-100, higher scores mean better outcome)
Clinical effectiveness (short-term) | 7 months post-injury
  Knee Injury and Osteoarthritis Outcome Score - Subscale Quality of Life (score between 0-100, higher scores mean better outcome)

SECONDARY OUTCOMES:
Prediction analysis to identify patient-specific factors that predict whether (or not) a patient will require delayed surgery | 36 months post-injury
  Dependent variable = whether or not delayed surgery is performed (binary event)
  Independent variables (candidate predictors):
  * Knee Injury and Osteoarthritis Outcome Score - Subscale Quality of Life at baseline
  * MRI findings at baseline scored with the modified ACLOAS (Anterior Cruciate Ligament OsteoArthritis Score)
  * Degree of hemarthrosis determined by MRI at baseline
  * Expectations regarding the effectiveness of physical therapy at baseline, measured with the illness perception questionnaire
  * Pre-injury activity level, measured with the Tegner Activity Score

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Smeets A, Ghafelzadeh Ahwaz F, Bogaerts S, Berger P, Peers K. Comparison of immediate versus optional delayed surgical repair for treatment of acute anterior cruciate ligament injury through a parallel, multicentric, pragmatic randomized controlled trial - IODA trial. BMC Sports Sci Med Rehabil. 2024 Jan 18;16(1):22. doi: 10.1186/s13102-024-00816-6. PMID 38238809